CLINICAL TRIAL: NCT01028079
Title: Placebo and Active Controlled, Double Dummy Phase III Study to Prove Efficacy of Aspirin (1000 mg Solid Dose) in Treatment of Acute Low Back Pain.
Brief Title: Placebo and Active Controlled, Double Dummy Study to Prove Efficacy of Aspirin in Treatment of Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11818
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Low Back Pain
Keywords: Back Pain; Acute low back pain
MeSH Terms: conditions — Low Back Pain; Back Pain | interventions — Aspirin; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 2 (Active Comparator)
  Interventions: Drug: Ibuprofen
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — Aspirin 1000 mg (solid dose caplet) to be given three times daily as for 2 consecutive days (48 hours), followed by Aspirin 1000 mg (solid dose caplet) to be taken as per need, but not more than three times daily for the following 3 days (72 hours). Total treatment period has not to exceed 5 days and total daily dose has not to exceed 3000 mg Aspirin.
  Arms: Arm 1
Drug: Ibuprofen — Ibuprofen 400 mg caplet to be given three times a day as for 2 consecutive days (48 hours), followed by ibuprofen 400 mg caplet to be given as per need, but not more than three times a day for the following 3 days (72 hours). Total treatment period has not to exceed 5 days and total daily dose has not to exceed 1200 mg ibuprofen.
  Arms: Arm 2
Drug: Placebo — Placebo (two placebos: Placebo Aspirin and Placebo Ibuprofen) to be given three times a day for a maximum of 5 consecutive days in the same regimen as for Experimental Drug and Active Comparator.
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine the efficacy and safety of 1000 mg Aspirin (the study medication) by comparing it to placebo (the control group without active substance) or 400 mg Ibuprofen (the control group with an active substance) in treating the symptoms of back pain. The study is designed to develop a treatment method against back pain which will have more advantages for patients than the methods that are currently available.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female, 18 to 70 years of age
* Body mass index ranging in-between 18 and 30 kg/m²
* Normal blood pressure
* Patients suffering from low back pain
* Low back pain, localized below the costal margin and above the inferior gluteal folds, either as acute low back pain, or as chronic or intermittent low back pain

Exclusion Criteria:

* Hypersensitivity to acetylsalicylic, salicylates, or other Non Steroidal Anti-inflammatory drugs
* Serious physical illness especially uncontrolled disorders of kidney, liver, lung, heart or brain function, neurological disorders or severe chronic or terminal disease
* Pregnancy or lactation period
* Abuse of alcohol or addictive substances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2005-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve of the baseline adjusted pain intensity curve over the initial 48 hours (AUC-PI0-48hours) after first dosing | 48 hours

SECONDARY OUTCOMES:
Total pain relief 6, 72, 96 and 120 hours after first dosing | 6, 72, 96 and 120 hours
Pain intensity relief over initial 6 hours | 6 hours
Pain intensity difference after 48, 72, 96 and 120 hours after first dosing | 48, 72, 96 and 120 hours
Overall efficacy after 48, 72, 96 and 120 hours after first dosing | 48, 72, 96 and 120 hours
Total dose used over 5 days | 5 days
Time till use of rescue medication | 5 days
Safety - assessment of adverse events | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Germany (7):
  - Bad Lippspringe
  - Beckum
  - Einbeck
  - Hamburg
  - Hanover
  - Künzing
  - Straßkirchen
- United Kingdom (3):
  - Fowey
  - Saltash
  - Sheffield